CLINICAL TRIAL: NCT03754517
Title: Finding the Latent Treponema Pallidum of Syphilis With Serofast Status
Brief Title: Finding the Latent Treponema Pallidum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: The reaseon of serofast
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2018-11

CONDITIONS: Syphilis
Keywords: syphilis; serofast
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — body fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Serofast status: The syphilitic patients who remain in a serologically positive state after therapy
  Interventions: Diagnostic Test: RPR Titer
- Untreated: untreated syphilis cases
  Interventions: Diagnostic Test: RPR Titer
- Serological cure: In the early syphilis patients, at 6 months following treatment, a serological cure was defined as either a negative RPR or ≥2 dilution (4-fold) decrease in the RPR titer.
  In the late syphilis patients, at 12 months following treatment, a serological cure was defined as either a negative RPR or ≥2 dilution (4-fold) decrease in the RPR titer.
  Interventions: Diagnostic Test: RPR Titer

INTERVENTIONS:
Diagnostic Test: RPR Titer — RPR titer; TPPA/FTA-ABS; Next-Generation Sequencing

SUMMARY:
Some syphilitic patients remain in a serologically positive state after the recommended therapy. Whether a serofast state could represent a persistent low-level infection by Treponema pallidum is still unknown. The possibility that persistent nontreponemal antibodies after treatment represent persistence of Treponema pallidum was raised by some investigators. The investigators use the Next-Generation Sequencing to test blood plasma, srum, cerebrospinal fluid, aqueous humor, lymph nodes, skin lesion, saliva, semen,milk of serofast patient and other positive and negative controls.

DETAILED DESCRIPTION:
Some syphilitic patients remain in a serologically positive state after the recommended therapy. Whether a serofast state could represent a persistent low-level infection by Treponema pallidum is still unknown. The possibility that persistent nontreponemal antibodies after treatment represent persistence of Treponema pallidum was raised by some investigators. The investigators use the Next-Generation Sequencing to test blood plasma, serum, cerebrospinal fluid, aqueous humor, lymph nodes, skin lesion, saliva, semen,milk of serofast patient and other positive and negative controls.

ELIGIBILITY:
Inclusion Criteria:

* All clinical diagnosis of syphilis cases

Exclusion Criteria:

* Auto-immune disease (such as SLE)
* Lyme disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All syphilis cases.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the reads of treponema pallidum | 30 days
  Using the Next-Generation Sequencing to test specific genome of treponema pallidum for syphilis

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- PekingUMCH, Beijing, China